CLINICAL TRIAL: NCT06180200
Title: Study of the in Vivo Expression of MU Opioid Receptors Using PET and the Selective Tracer [C-11] Carfentanil in Normal Weight and Obese Subjects
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: CARF-2
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Nuclear Medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET for the analysis of mu opioid receptor expression. — PET for the analysis of the expression of mu opioid receptors and to directly measure the distribution of the receptors and enzyme reuptake sites at the brain level.

SUMMARY:
Positron emission tomography (PET) is a nuclear medicine technique that allows the measurement, in vivo in humans, with a non-invasive method, of the regional distribution of substances marked with positron emission isotopes such as C-11, in different districts bodily. Using this method it is therefore possible to directly measure at the level of the brain the distribution of receptors, enzymes, reuptake sites, as well as their interaction with various classes of drugs and the related modifications that may be present during the pathology.

The evaluation of the endogenous opiate receptor system will be implemented by comparing the in vivo binding maps of 11C carfentanil in the two groups of subjects under examination (normal weight, NOR and obese, OB, based on body mass index, BMI); in fact, experimental data deriving from previous studies support the hypothesis that the basis of obesity and incorrect eating behaviors is a dysregulation of the endogenous ligand-mu opioid receptor interaction. The comparison of the data deriving from the analysis of the PET exams performed on the two groups of subjects will therefore allow us to evaluate the alterations of the opioid system possibly present in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 40 years;
* structured sports activity < 2 hours per week

Exclusion Criteria:

* drug allergy;
* clinical evidence of neuropsychiatric pathologies.

Ages: 18 Years to 40 Years | Sex: Male
Age Groups: Adult
Study Population: For the study, 10 normal male subjects and 10 obese subjects not affected by mental or physical pathological alterations will be recruited.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2004-10-22 (Actual); Primary Completion 2007-12-01 (Actual); Study Completion 2007-12-01 (Actual)

PRIMARY OUTCOMES:
PET with 11C CARFENTANIL for the analysis of the expression of mu opioid receptors. | 3 years
  Study of the expression of mu opioid receptors in normal weight and obese subjects

IPD SHARING:
Plan to Share IPD: No